CLINICAL TRIAL: NCT00854568
Title: A Randomized Phase III Study Comparing CHOP Versus CEOP-induced Cardiotoxicity in Patients With Aggressive B-cell Lymphoma
Brief Title: Comparison Study of Doxorubicin Versus Epirubicin-induced Cardiotoxicity in Patients With DLBCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 09-01
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Lymphoma
Keywords: B-cell lymphoma; CHOP; CEOP; Cardiotoxicity
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Cardiotoxicity | interventions — CEOP protocol 1; VAP-cyclo protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CEOP regimen (Experimental): CEOP regimen
  Interventions: Drug: CEOP regimen
- CHOP regimen (Active Comparator): CHOP regimen
  Interventions: Drug: CHOP regimen

INTERVENTIONS:
Drug: CEOP regimen — cyclophosphamide 750mg/m2 IV day 1 epirubicin 70mg/m2 IV day 1 vincristine 1.4mg/m2 IV day1 (maximum: 2mg) prednisone 50mg PO days 1~5 twice per day Or combined with rituximab 375mg/m2 IV day 0
  Other Names: CEOP
  Arms: CEOP regimen
Drug: CHOP regimen — cyclophosphamide 750mg/m2 IV day 1 doxorubicin 50mg/m2 IV day 1 vincristine 1.4mg/m2 IV day1 (maximum: 2mg) prednisone 50mg PO days 1~5 twice per day Or combined with rituximab 375mg/m2 IV day 0
  Other Names: CHOP
  Arms: CHOP regimen

SUMMARY:
The aim of this study is to compare CHOP versus CEOP-induced cardiotoxicity in patients with aggressive B-cell lymphoma. The hypothesis is epirubicin is associated with less cardiotoxicity without compromising the efficacy.

DETAILED DESCRIPTION:
The doxorucin-containing regimen (CHOP) and epirubicin-containing regimen (CEOP) are both frequently used in patients with aggress B-cell lymphoma in out institution. According to a Cochrane meta-analysis, epirubicin is less cardiotoxic than doxorubicin on a mg per mg basis. However, compared with 50mg/m2 of doxorubicin in CHOP, epirubicin was usually used at a higher dose (70mg/m2) to treat non-Hodgkin's lymphoma (NHL). Because of the correlation between cumulative dose and risk of cardiotoxicity, it is reasonable to speculate that CEOP (70mg/m2) has less cardiotoxicity than CHOP (50mg/m2) when both regimens are administered with similar cycles.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated aggressive B-cell lymphoma
* Age range 18-75 years old
* ECOG performance status 0-2
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

* Previous serious cardiac disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity (Class III or IV cardiotoxicity according to New York Heart Association (NYHA) Classification or LVEF abnormality [< 50% or a decrease in absolute LVEF ≥ 10%) by post-treatment RNA]) | 18 weeks

SECONDARY OUTCOMES:
Objective response rate | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China